CLINICAL TRIAL: NCT05086744
Title: An Open-label, Multi-center, Phase 2 Basket Study to Assess Efficacy, Safety and Pharmacokinetics of Iptacopan (LNP023) in Participants With Autoimmune Benign Hematological Disorders
Brief Title: Basket Study to Assess Efficacy, Safety and PK of Iptacopan (LNP023) in Autoimmune Benign Hematological Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023L12201; 2021-002039-40 (EudraCT Number)
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Immune Thrombocytopenia (ITP); Cold Agglutinin Disease (CAD)
Keywords: LNP023; Iptacopan; Immune thrombocytopenia; Cold agglutinin disease; Autoimmune benign hematological disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune | interventions — iptacopan; Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: This is a basket study with different Cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iptacopan 200 mg BID (Experimental): Iptacopan 200 mg twice daily (BID) in participants with primary ITP and primary CAD
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Iptacopan 200 mg BID given orally (capsule)
  Other Names: Investigational new drug; company code: LNP023

SUMMARY:
The main purpose of this study was to evaluate the efficacy and safety of iptacopan in participants with autoimmune benign hematological disorders such as primary immune thrombocytopenia and primary cold agglutinin disease.

DETAILED DESCRIPTION:
This was an open-label, single-arm (within each cohort), multi-center, non-confirmatory basket study to assess the efficacy, safety and pharmacokinetics of iptacopan in participants with autoimmune benign hematological disorders. The study was set up as a basket study to allow inclusion of new cohorts (indications). The study included 2 cohorts: primary immune thrombocytopenia (ITP) and primary cold agglutinin disease (CAD). Participants in Cohort 1 (ITP) were stratified in two groups according to high/low complement activation (i.e., based on sC5b-9 level at screening). No additional cohorts were added during the study.

The study consisted of a screening period, a 12-week treatment period (Part A), a washout (for responders)/follow-up (for non-responders) period after Part A, and, for responders only, an additional treatment extension period for up to 24 months (Part B). Non-responders who had signs of clinical benefit according to the Investigator's assessment could also continue treatment with iptacopan in Part B. The washout period prior to the start of part B lasted up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Written informed consent
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infections was required and vaccination against Haemophilus influenzae infection is recommended prior to the start of treatment.
* Weight of at least 35 kg

Cohort 1 specific inclusion criteria:

* Participants with a diagnosis of persistent or chronic primary ITP
* Participants must have received at least 1 unique prior therapy administered with the intention to treat ITP
* Sustained thrombocytopenia

Cohort 2 specific inclusion criteria:

* Participants with a diagnosis of primary CAD
* Participants must have received at least 1 unique prior therapy administered with the intention to treat CAD
* Laboratory evidence of ongoing hemolysis
* Sustained anemia

Exclusion Criteria:

All cohorts:

* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations
* Past or concomitant use of medications prohibited by the protocol
* Known or suspected hereditary or acquired complement deficiency
* History of primary or secondary immunodeficiency, including a positive HIV test result
* Chronic infection with Hepatitis B or C virus
* History of recurrent invasive infections caused by encapsulated organisms, including Neisseria meningitidis, Streptococcus pneumoniae, or Haemophilus influenzae
* Presence or suspicion of any active infection within 14 days prior to first study drug administration.
* Any medical condition deemed likely to interfere with the participant's participation in the study
* Any malignant disease diagnosed within the past 5 years, with the exception of localized non-melanoma skin cancer, in situ cervical cancer, or, for CAD, a low-grade lymphoproliferative disorder.
* History of bone marrow/hematopoietic stem cell or solid organ transplantation.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of investigational drug and for 1 week after last iptacopan dose
* Active severe bleeding or history of intracranial hemorrhage.
* Liver disease, or liver injury as indicated by abnormal liver function tests.
* Severe concurrent comorbidities of unstable medical conditions.

Cohort 1 specific exclusion criteria:

* Secondary ITP, as may arise in the setting of certain autoimmune disorders, immunodeficiency syndromes, infections, malignancies, and drug treatments
* No ITP-directed background therapy permitted, with the exception of either a thrombopoietin receptor agonist or low-dose corticosteroid, as long as stable dosage for at least 4 weeks prior to first iptacopan dose
* Abnormal coagulation screening labs

Cohort 2 specific exclusion criteria:

* Secondary cold agglutinin syndrome, as may arise in the setting of certain infections, autoimmune disorders, and malignancies (with the exception of a low-grade lymphoproliferative disorder)
* No CAD-directed background therapy permitted

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient level data and supporting clinical documents from applicable studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Roth A, Barcellini W, Ademokun C, Jang J, Lozano ML, Ferreiras DV, Pascual-Izquierdo C, Chitnis S, Matviykiv S, Vitaliti A, Chen C, Katsanou V, Chawla R, Al-Samkari H. Iptacopan for Immune Thrombocytopenia and Cold Agglutinin Disease: A Global Phase 2 Basket Clinical Trial. Am J Hematol. 2026 Feb;101(2):242-254. doi: 10.1002/ajh.70147. Epub 2025 Dec 9. PMID 41366634
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 8 investigative sites in 6 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations had to be completed within 8 weeks prior to the first dose of study treatment. The treatment period started on Day 1 of Part A.
Groups:
- Cohort 1 (ITP): Iptacopan 200 mg twice daily (b.i.d.) in participants with primary immune thrombocytopenia (ITP)
- Cohort 2 (CAD): Iptacopan 200 mg twice daily (b.i.d.) in participants with primary cold agglutinin disease (CAD)
Period: Part A
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Started | 9 | 10
PD Analysis Set (All participants who received any study drug and with no protocol deviations with relevant impact on pharmacodynamics (PD) data) | 8 | 10
ITP - sC5b-9 Low (Participants with primary ITP and low complement activation (low sC5b-9 levels)) | 5 | 0
ITP - sC5b-9 High (Participants with primary ITP and high complement activation (high sC5b-9 levels)) | 4 | 0
Completed | 4 | 9
Not Completed | 5 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol deviation | 1 | 0
Not completed — Subject decision | 1 | 0
Period: Part B
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Started | 1 | 8
ITP - sC5b-9 High (Participants with primary ITP and high complement activation (high sC5b-9 levels)) | 1 | 0
ITP - sC5b-9 Low (Participants with primary ITP and low complement activation (low sC5b-9 levels)) | 0 | 0
Completed | 0 | 0
Not Completed | 1 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study terminated by sponsor | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD) | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (20.77) | 66.7 (10.01) | 56.1 (19.36)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 7 | 5 | 12
  65 - <85 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 4 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 3
  White | 6 | 10 | 16
Platelets [Mean (Standard Deviation); unit: platelets*10^9/liter] — Platelet count in blood at baseline for participants in Cohort 1 Population: Study specific characteristic for participants in Cohort 1 only.
  platelets*10^9/liter
    number analyzed (Participants) | 9 | 0 | 9
    (all) | 14.6 (10.53) |  | 14.6 (10.53)
Hemoglobin [Mean (Standard Deviation); unit: gram/liter] — Hemoglobin in blood at baseline for participants in Cohort 2 Population: Study specific characteristic for participants in Cohort 2 only.
  gram/liter
    number analyzed (Participants) | 0 | 10 | 10
    (all) |  | 86.7 (9.06) | 86.7 (9.06)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 (ITP): Number of Participants With a Clinically Meaningful Response
Description: A study participant with ITP was considered a responder if all the below criteria were met:
  1. Platelet count of ≥50 k/μL sustained for at least 2 consecutive weeks during the main, 12-week treatment part
  2. Absence of rescue therapy or prohibited medications to treat ITP
  3. Lack of treatment discontinuation
Time Frame: Up to 12 weeks (Part A)
Population: Participants from Cohort 1 in the Pharmacodynamic (PD) analysis set. Results are presented by sC5b-9 stratification group (sC5b-9 high and sC5b-9 low) and overall.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (ITP) - sC5b-9 High: Iptacopan 200 mg b.i.d. in participants with primary ITP and high complement activation (i.e., high sC5b-9 levels)
- Cohort 1 (ITP) - sC5b-9 Low: Iptacopan 200 mg b.i.d. in participants with primary ITP and low complement activation (i.e., low sC5b-9 levels)
Arm/Group | Cohort 1 (ITP) - sC5b-9 High | Cohort 1 (ITP) - sC5b-9 Low | Cohort 1 (ITP)
Number analyzed (Participants) | 3 | 5 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Cohort 2 (CAD): Number of Participants With a Clinically Meaningful Response
Description: A study participant with CAD was considered a responder if all the below criteria were met:
  1. Hemoglobin level increase of ≥1.5 g/dL above baseline sustained for at least 2 consecutive weeks during the main, 12-week treatment part
  2. Absence of rescue therapy or prohibited medications to treat CAD
  3. Lack of treatment discontinuation
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 10
Participants | 5

3. Secondary Outcome: Cohort 1 (ITP): Time to First Platelet Count ≥50 k/μL
Description: The first time that a participant had a platelet count ≥50 k/μL after first dose of study treatment. Time to the first response was assessed for responders only.
Time Frame: Up to 12 weeks (Part A)
Population: Participants from Cohort 1 in the Pharmacodynamic (PD) analysis set who were responders. Results are presented by sC5b-9 stratification group (sC5b-9 high and sC5b-9 low) and overall.
Arm/Group | Cohort 1 (ITP) - sC5b-9 High | Cohort 1 (ITP) - sC5b-9 Low | Cohort 1 (ITP)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Cohort 2 (CAD): Time to First Hemoglobin Level ≥1.5 g/dL Above Baseline
Description: The first time that a participant had a hemoglobin level ≥1.5 g/dL above baseline after first dose of study treatment. Time to the first response was assessed for responders only.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set who were responders.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 5
days | 29.0 [23 to 63]

5. Secondary Outcome: Cohort 1 (ITP): Duration of Time During Which Platelet Count Remains ≥50 k/μL Without the Use of Rescue Therapy
Description: The duration of response corresponds to the duration of time during which a participant's platelet count remains ≥50 k/μL without the use of rescue therapy. The duration of response was considered as cumulative if there were non-continuous periods of response. Duration of response was analyzed for responders only.
Time Frame: Up to 12 weeks (Part A)
Population: as for outcome 3
Arm/Group | Cohort 1 (ITP) - sC5b-9 High | Cohort 1 (ITP) - sC5b-9 Low | Cohort 1 (ITP)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Cohort 2 (CAD): Duration of Time During Which Hemoglobin Level Remains ≥1.5 g/dL Above Baseline Without the Use of Rescue Therapy
Description: The duration of response corresponds to the duration of time during which a participant's hemoglobin level remained ≥1.5 g/dL above baseline without the use of rescue therapy. The duration of response was considered as cumulative if there were non-continuous periods of response. Duration of response was analyzed for responders only.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set who were responders.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 5
days | 56.0 [28 to 63]

7. Secondary Outcome: Cohort 1 (ITP): Magnitude of Platelet Count Increase From Baseline
Description: The magnitude of increase in platelet count compared to baseline was derived for each participant at each visit and time point. Best response across all visits is presented (highest value).
  The following categories were used: absolute platelet counts increase <50, ≥50 and <100, ≥100 and <150, and ≥150 k/uL.
  This endpoint is only applicable to participants without rescue therapy in the treatment period.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 1 in the Pharmacodynamic (PD) analysis set who did not use rescue therapy in the treatment period of Part A. Results are presented by sC5b-9 stratification group (sC5b-9 high and sC5b-9 low) and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (ITP) - sC5b-9 High | Cohort 1 (ITP) - sC5b-9 Low | Cohort 1 (ITP)
Number analyzed (Participants) | 1 | 2 | 3
Participants
  Absolute platelet counts increase <50 k/uL | 1 | 2 | 3
  Absolute platelet counts increase >=50 k/uL and <100 k/uL | 0 | 0 | 0
  Absolute platelet counts increase >=100 k/uL and <150 k/uL | 0 | 0 | 0
  Absolute platelet counts increase >=150 k/uL | 0 | 0 | 0

8. Secondary Outcome: Cohort 2 (CAD): Magnitude of Hemoglobin Increase From Baseline
Description: The magnitude of increase in hemoglobin level compared to baseline was derived for each participant at each visit and time point. Best response across all visits is presented (highest value).
  The following categories were used: Hb increase from baseline by <1, ≥1 and <1.5, ≥1.5 and <2, and ≥2 g/dL.
  This endpoint is only applicable to participants without rescue therapy in the treatment period.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set who did not use rescue therapy in the treatment period of Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 9
Participants
  Hb increase by <1.0 g/dL | 2
  Hb increase by >=1.0 g/dL and <1.5 g/dL | 1
  Hb increase by =>1.5 g/dL and <2 g/dL | 2
  Hb increase by =>2 g/dL | 4

9. Secondary Outcome: Cohort 1 (ITP): Need for Rescue Therapy During Part A
Description: Rescue therapy was defined as any therapy with ITP indication that started on or after Day 1.
  Rescue therapy, if indicated, could be initiated at the Investigator's discretion. From Day 1 onwards, if rescue therapy was needed before response criteria were met, the participant was treated as a non-responder. Conversely, use of rescue therapy after the primary endpoint was met, would not impact the response status with respect to that endpoint.
  For ITP, rescue therapy generally consisted of corticosteroids, intravenous immunoglobulins or anti-Rho(D) immunoglobulin and may had been indicated in case of worsening thrombocytopenia and/or signs or symptoms of bleeding.
Time Frame: Up to 12 weeks (Part A)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (ITP) - sC5b-9 High | Cohort 1 (ITP) - sC5b-9 Low | Cohort 1 (ITP)
Number analyzed (Participants) | 3 | 5 | 8
Participants
  No | 1 | 2 | 3
  Yes | 2 | 3 | 5

10. Secondary Outcome: Cohort 2 (CAD): Need for Rescue Therapy During Part A
Description: Rescue therapy was defined as any therapy with CAD indication that started on or after Day 1.
  Rescue therapy, if indicated, could be initiated at the Investigator's discretion. From Day 1 onwards, if rescue therapy was needed before response criteria were met, the participant was treated as a non-responder. Conversely, use of rescue therapy after the primary endpoint was met, would not impact the response status with respect to that endpoint.
  For CAD, rescue therapy generally consisted of plasmapheresis, intravenous immunoglobulins (IVIG) and/or red blood cell transfusions and may had been indicated in case of worsening anemia and/or critical hemolysis.
Time Frame: Up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 10
Participants
  No | 9
  Yes | 1

11. Secondary Outcome: Cohort 2 (CAD): Change From Baseline in Lactate Dehydrogenase (LDH)
Description: LDH was measured in serum samples to assess the effect of treatment with iptacopan on relevant disease biomarkers.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: Participants from Cohort 2 in the PD analysis set with an available value for the outcome measure at both baseline and end of treatment in Part A.
Measure: Mean (Standard Deviation); unit: Units/liter (U/L)
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 6
Units/liter (U/L) | -277.83 (88.966)

12. Secondary Outcome: Cohort 2 (CAD): Change From Baseline in Total Bilirubin
Description: Total bilirubin was measured in serum samples to assess the effect of treatment with iptacopan on relevant disease biomarkers.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micromole/liter (μmol/L)
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 8
micromole/liter (μmol/L) | -15.63 (12.979)

13. Secondary Outcome: Cohort 2 (CAD): Change From Baseline in Reticulocyte Count
Description: Reticulocyte count was measured in blood samples to assess the effect of treatment with iptacopan on relevant disease biomarkers.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: reticulocytes * 10^9/liter
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 8
reticulocytes * 10^9/liter | -37.45 (17.205)

14. Secondary Outcome: Cohort 2 (CAD): Change From Baseline in Haptoglobin
Description: Haptoglobin was measured in serum or plasma samples to assess the effect of treatment with iptacopan on relevant disease biomarkers.
Time Frame: Baseline, up to 12 weeks (Part A)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: gram/liter (g/L)
Arm/Group | Cohort 2 (CAD)
Number analyzed (Participants) | 9
gram/liter (g/L) | 0.12 (0.236)

15. Secondary Outcome: Cohort 1 and 2: Number of Participants With AEs and SAEs During the On-treatment Period in Part A and B
Description: Number of participants with AEs (any adverse events regardless of seriousness) and serious adverse events (SAEs), including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. For CTCAE v5.0, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The on-treatment period is defined from the day of first administration of study drug up to 7 days after the last administration of study drug.
Time Frame: From first dose of study treatment to 7 days after last dose, up to approximately 43 weeks (Cohort 1) and 103 weeks (Cohort 2)
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Number analyzed (Participants) | 9 | 10
Participants
  AEs | 7 | 9
  Treatment-related AEs | 2 | 3
  Severe AEs | 1 | 0
  Treatment-related severe AEs | 1 | 0
  SAEs | 0 | 1
  Treatment-related SAEs | 0 | 0
  Fatal SAEs | 0 | 0
  Treatment-related fatal SAEs | 0 | 0

16. Secondary Outcome: Cohort 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Iptacopan
Description: Pharmacokinetic (PK) parameters were calculated based on iptacopan plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Pre-dose, 0.5, 2, 4 and 6 hours after iptacopan administration on Day 15 and Day 57 of Part A
Population: Participants in the PK analysis set (PAS) who had an available value for the outcome measure on the assessed study day. PAS consisted of all participants with at least one available valid PK concentration measurement, who received any study drug and with no protocol deviations or AEs which may have impacted iptacopan's PK.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Number analyzed (Participants) | 7 | 9
ng/mL
  Day 15: number analyzed (Participants) | 7 | 8
  Day 15 | 3190.0 (465.00) | 4800.0 (838.00)
  Day 57: number analyzed (Participants) | 3 | 9
  Day 57 | 2940.0 (1020.00) | 4420.0 (1300.00)

17. Secondary Outcome: Cohort 1 and 2: Time to Maximum Observed Plasma Concentration (Tmax) of Iptacopan
Description: PK parameters were calculated based on iptacopan plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) observed concentration following a dose. Actual sampling times were considered for the calculation of PK parameters.
Time Frame: Pre-dose, 0.5, 2, 4 and 6 hours after iptacopan administration on Day 15 and Day 57 of Part A
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Number analyzed (Participants) | 7 | 9
hours
  Day 15: number analyzed (Participants) | 7 | 8
  Day 15 | 2 [0.75 to 5.15] | 1 [1 to 2]
  Day 57: number analyzed (Participants) | 2 | 9
  Day 57 | 2 [2 to 2] | 1.97 [1 to 2]

18. Secondary Outcome: Cohort 1 and 2: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Iptacopan
Description: PK parameters were calculated based on iptacopan plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve (AUC) calculation.
Time Frame: Pre-dose, 0.5, 2, 4 and 6 hours after iptacopan administration on Day 15 and Day 57 of Part A
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Number analyzed (Participants) | 7 | 9
hr*ng/mL
  Day 15: number analyzed (Participants) | 7 | 8
  Day 15 | 24200.0 (6110.00) | 31100.0 (5830.00)
  Day 57: number analyzed (Participants) | 3 | 9
  Day 57 | 21300.0 (5280.00) | 28200.0 (6880.00)

19. Secondary Outcome: Cohort 1 and 2: Trough Plasma Concentration (Ctrough) of Iptacopan
Description: Ctrough is defined as the concentration reached immediately before the next dose is administered. All drug concentrations below the lower limit of quantification were treated as zero for the calculation of PK parameters.
Time Frame: Pre-dose on Day 15, 29 and 57 of Part A
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD)
Number analyzed (Participants) | 8 | 9
ng/mL
  Day 15 | 1670.0 (1320.00) | 1980.0 (1720.00)
  Day 29: number analyzed (Participants) | 6 | 7
  Day 29 | 1670.0 (927.00) | 1330.0 (337.00)
  Day 57: number analyzed (Participants) | 5 | 9
  Day 57 | 1680.0 (758.00) | 1410.0 (320.00)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to 30 days after last dose, up to approximately 46 weeks (Cohort 1) and 106 weeks (Cohort 2)
Groups:
- All Patients: All patients in the study
Arm/Group | Cohort 1 (ITP) | Cohort 2 (CAD) | All Patients
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10 | 2/19
Other Adverse Events (participants affected / at risk) | 7/9 | 9/10 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (ITP) (N=9) | Cohort 2 (CAD) (N=10) | All Patients (N=19)
Blood creatinine increased (Investigations) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (ITP) (N=9) | Cohort 2 (CAD) (N=10) | All Patients (N=19)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 3 | 3
Pyrexia (General disorders) | 0 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1
Fungal foot infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood iron increased (Investigations) | 0 | 1 | 1
Reverse tri-iodothyronine increased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 5
Depressed mood (Psychiatric disorders) | 0 | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT05086744/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05086744/SAP_001.pdf